CLINICAL TRIAL: NCT02406638
Title: Pelvic Floor 3D Ultrasound of Women Who Underwent TVT-R, TVT-O, TVT-S Surgery at Three Years Follow-up
Brief Title: Pelvic Floor 3D USG Three Years After Mid-urethral Slings ( TVT-R, TVT-O, TVT-S)
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, PhD, Federal University of São Paulo
Other Study IDs: CAAE12805313800005505
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Urinary Incontinence; Postoperative Period
Keywords: 3D Pelvic floor USG; Mid-Urethral Sling; TVT; TVT-O; TVT-S
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- TVT Group: Women who underwent to stress urinary incontinence surgery using Gynecare TVT 3 years before clinical and 3D pelvic floor ultrasound evaluation.
  Interventions: Other: 3D pelvic floor ultrasound
- TVT-O Group: Women who underwent to stress urinary incontinence surgery using Gynecare TVT Obturator System, inside-out approach, 3 years before clinical and 3D pelvic floor ultrasound evaluation.
  Interventions: Other: 3D pelvic floor ultrasound
- TVT-S Group: Women who underwent to stress urinary incontinence surgery using GynecareTVT-Secur System, in "U" approach, 3 years before clinical and 3D pelvic floor ultrasound evaluation.
  Interventions: Other: 3D pelvic floor ultrasound

INTERVENTIONS:
Other: 3D pelvic floor ultrasound — Pelvic Floor 3D Ultrasound Clinical evaluation with pad-test, stress test and questionnaires of symptoms and quality of life

SUMMARY:
Compare through 3D USG the tape spatial orientation, in three different techniques of insertion of mid-urethral synthetic sling, correlating USG findings to postoperative results in an average of three years follow-up.

Methods: This is a transversal study of a cohort women surgically treated for stress urinary incontinence by retropubic sling (TVT-R), transobturator sling (TVT-O) or single-incision sling (TVT-S). The clinical and USG evaluation were performed at the same medical visit, from April 2013 to June 2014, .

DETAILED DESCRIPTION:
Introduction: The three dimensional ultrasonography (3D USG) provides a clear spatial orientation of polypropylene tape and can help clarify the pathogenesis of bladder dysfunction after a TVT procedure. Thus, the USG in urogynecology postoperative has shown an increasing role in monitoring surgically treated patients and specially in complications such as urinary retention and urinary disorders.

Objective: Compare through 3D USG the tape spatial orientation, in three different techniques of insertion of mid-urethral synthetic sling, correlating USG findings to postoperative results in an average of three years follow-up.

Methods: This is a transversal study of a cohort of women surgically treated for stress urinary incontinence by retropubic sling (TVT-R), transobturator sling (TVT-O) or single-incision sling (TVT-S). The surgeries occurred from May 2009 to December 2011. Were eligible for the study 158 patients. The clinical and USG evaluation were performed at the same medical visit, from April 2013 to June 2014, after local ethics committee approval and signature of informed consent. The objective cure rates were evaluated by negative pad-test and stress test. The subjective cure rate and urgency symptoms were accessed by questionnaires. The subjective cure was defined as absence of reports of stress urinary leakage.

The USG evaluation was performed using General Electric Voluson 730 expert systems with 8 - 4 Mhz volume transducers with an 85-degree acquisition angle. The exams were performed with patient in supine position with hip flexed and using slightly abduced, after voiding. The US transducer was placed on the perineum in the midsagittal position and volumes were obtained at rest, at maximum Valsalva, and perineal contraction. Moved mode rendering for OMNINI View plan as previous described.The volumes datasets were analyzed offline by of the authors. They were blinded and the average values were considered.

The urethral length and the location of the sling, measured by the distance between bladder neck and the tape (CF), were assessed in midsagittal plane. The tape angle in relation to the urethra were assessed in OMINI VIEW plan.

Statistical analysis was performed using student t, ANOVA and Tukey-test. P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent surgical treatment for stress urinary incontinence using TVT, TVT-O and TVT-Secur, in a period of 2 to 4 years before the USG evaluation
* Informed consent signed

Exclusion Criteria:

* Patients who underwent to more than one surgery for urinary incontinence using polypropylene tape
* Ultrasound images that would not allow adequate visualization of the tape

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who underwent stress urinary incontinence surgery with synthetic midurethral sling, by different approaches ( TVT, TVT-O and TVT-Secur) in a period of 2 to 4 years before clinical and 3D USG evaluation
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Determination of the tape spatial position ( angle between tape arms surrounding urethra measured in grades) in three different techniques of insertion of midurethral synthetic sling (TVT, TVT-O, TVT-S) | evaluation will occur in 1 day, 3 years after surgery
  Measured of the angle between tape arms surrounding urethra (in grades) in the three different suburethral tapes measured by 3D USG at rest Valsalva and pelvic floor contraction

SECONDARY OUTCOMES:
Correlation between the suburethral tape spatial positon and objective cure rate | evaluation will occur in 1 day, 3 years after surgery
  Correlation between the tape spatial position measured by 3D USG and objective cure rates, accessed by stress test and pad-test
Correlation between the suburethral tape spatial positon and subjective cure rate | evaluation will occur in 1 day, 3 years after surgery
  Correlation between the tape spatial position measured by 3D USG and subjective cure, accessed by scale of symptoms of King's Health Questionnaire
Correlation between the suburethral tape spatial positon and urge-symptoms | evaluation will occur in 1 day, 3 years after surgery
  Correlation between the tape spatial position measured by 3D USG and urge-symptoms, accessed by scale of symptoms of King's Health Questionnaire
Determination of the tape position, distance between the tape and vesical neck (measured in mm) in three different techniques of insertion of midurethral synthetic sling (TVT, TVT-O, TVT-S) | evaluation will occur in 1 day, 3 years after surgery
  Measured of the distance between the tape and vesical neck, in mm, of the three different suburethral tapes measured by 3D USG at rest Valsalva and pelvic floor contraction.
Determination of the tape position, relation between urethral length and distance between tape and vesical neck (measured in mm) in three different techniques of insertion of midurethral synthetic sling (TVT, TVT-O, TVT-S) | evaluation will occur in 1 day, 3 years after surgery
  Relation between the measured of urethral length (mm) and the distance between the tape and vesical neck( in mm), measured by 3D USG at rest Valsalva and pelvic floor contraction of the three different suburethral tapes, in order to determine if they remain in the midurethra.

CONTACTS AND LOCATIONS:
Overall Officials: Claudinei A Rodrigues, MD, Principal Investigator — Federal University of São Paulo; Zsuzsanna IK Jármy-di-Bella, PhD, Study Chair — Federal University of São Paulo; Ana Maria HM Bianchi-Ferraro, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo - Unifesp, São Paulo, São Paulo, Brazil